CLINICAL TRIAL: NCT05039307
Title: Prevention of Type 2 Diabetes and Gestational Diabetes Among Women of Reproductive Age in Kisantu, Democratic Republic of Congo
Brief Title: Prevention of Type 2 Diabetes and Gestational Diabetes Among Women in Kisantu, Democratic Republic of Congo
Acronym: KIS-Antwerp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Memisa, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1482/21
Record Dates: First submitted 2021-08-19; First posted 2021-09-09 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 2; Gestational Diabetes
Keywords: Prevention; Type 2 diabetes; Gestational diabetes; Women of reproductive age; Healthy lifestyle; Democratic Republic of the Congo
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: A cluster randomized controlled trial (cRCT) with a hierarchical design will be conducted whereby 2 groups of 3 healthcare centers (in total 6 healthcare centers) will be randomized to an intervention group or comparison group.
Masking Description: Masking is not possible due to the nature of this research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Educational and motivational strategy) (Experimental): The intervention group will be provided with a multi-component intervention entailing the following components distributed over the 24-months study: 4 individualized education sessions at the household, 4 group activities (2 group education sessions and 2 physical activity sessions) at the healthcare center, and 4 focus groups at the healthcare center as well. The motivational components of goal setting and the use of a pedometer will be incorporated in the individualized education sessions. Moreover, community activities will be incorporated in the second year of the study after exploring whether the activities are feasible and acceptable by the community. The topics covered by the intervention are healthy diet, physical activity, weight control strategies and knowledge and awareness of T2DM and GDM. Additionally, at baseline participants will be provided with a healthy lifestyle brochure with general recommendations.
  Interventions: Behavioral: Educational and motivational strategy
- Comparison group (Basic educational strategy) (No Intervention): The comparison group will be limited to receive the healthy lifestyle brochure with general recommendations at baseline only.

INTERVENTIONS:
Behavioral: Educational and motivational strategy — The intervention will focus on the following topics A) Healthy diet: food pyramid, a healthy plate distribution, type of carbohydrates and fats, healthy cooking techniques and healthy oils. B) Physical activity: definition, types of physical activity, advantages and benefits, examples, active physical activity sessions. C) Weight control: strategies, benefits and healthy weight gain during pregnancy. D) Knowledge and awareness of T2DM and GDM: definition, prevention, management and complications. These topics will be delivered through individualized education, group sessions and focus groups. Participants will be provided with printed material at baseline and also during the individual education sessions at the household containing a brief summary of the topics covered. The motivational components of goal setting and the use of a pedometer will be incorporated explained during the individual education sessions. The intervention will be primarily delivered by trained peer educators.
  Arms: Intervention group (Educational and motivational strategy)

SUMMARY:
This study aims to develop and implement a long-term program focused on the prevention of type 2 diabetes Mellitus (T2DM) and gestational diabetes mellitus (GDM) in women of reproductive age through lifestyle modification. This is a cluster-randomized trial whereby 6 health centers across Kisantu, Democratic Republic of Congo (DRC) will be randomized to an intervention group (3 health centers) or a comparison group (3 health centers). The intervention group will be provided with a preventive program based on educational + motivational strategies when the comparison group will be limited to an educational strategy only. This study will last 24 months and is limited to women of reproductive age (18-49 years), pregnant and non-pregnant. Evaluation of this research will use mixed longitudinal analyses for healthy lifestyle adherence, anthropometric and clinical indicators, diet quality, and physical activity. Expected results of this study for women of reproductive age include the prevention of T2DM and GDM through the acquisition of healthy lifestyle behavior, reaching and maintaining an optimal weight, blood pressure and glycemia, and adhere to the weight gain recommendations during pregnancy. Other expected achievements encompass improvements in the usability of data capturing systems, expand knowledge among health care providers on effective strategies for T2DM and GDM prevention and improve the technique and precision of measurements concerning health visits among health care providers, among others.

DETAILED DESCRIPTION:
Background: As the obesity epidemic continues to rise, it is expected that rates of T2DM and GDM will be also increasing among women in Sub-Saharan Africa (SSA). Women of reproductive age are a particularly vulnerable group, and there is a need for preventive programs addressing the incidence of obesity, T2DM, and GDM.

Objective: This study aims to develop, implement, and evaluate a long-term program (KIS-Antwerp) focused on the prevention of T2DM and GDM in women through a healthy lifestyle promotion.

Methods: The study will take place in 6 healthcare centers across Kisantu, DRC, and will be limited to women of reproductive age (18-49 years) irrespectively of pregnancy status. KIS-Antwerp will be implemented and evaluated using a matched cluster randomized controlled trial where the 6 healthcare will be randomized into an intervention group and a comparison group. The duration of the present study is 24 months. A total of 144 participants per arm is necessary to detect a 12% change in the primary outcome with a level of significance of 0.05, power >80%, and considering a 20% loss of follow-up. The intervention group will be provided with a preventive intervention program based on educational + motivational strategies including the following intervention program components: Individualized education, group education, physical activity sessions, setting goals, and usage of a pedometer. The comparison group will be limited to a basic educational strategy only (basic individual education). Participants will be followed up for 24 months and measurements will be assessed every 6-months period.

Statistical methods: Demographic characteristics will be reported as measures of central tendency for continuous outcomes and frequency distribution and percentages for binary/categorical data. Consequently, demographic data will be explored for differences at baseline by comparing and testing means. After the termination of the study, the primary and secondary outcomes will be evaluated for normality by the Kolmogorov-Simonov test and visual inspection of histograms. For the primary ordinal outcome, the impact of the intervention program between baseline and follow up of the 2 groups (intervention and comparison group) will be assessed by using linear mixed models for repeated measurements.

Safety: This study imposes a low risk for the participants as the intervention program compromises a lifestyle modification through education and motivational strategies and the measurements to be taken are non-invasive, with the exception of blood glucose assessment by blood sampling using a finger prick. For this measurement, guidelines with all the necessary steps and equipment will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant or (first trimester) pregnant women
* Women of reproductive age (18-49 years old)
* Without a previous diagnosis of type 1 diabetes or T2DM (confirmed by a random glucose test)

Exclusion Criteria:

* Pregnant women with active gestational diabetes
* Adult males, and children and adolescents <18 years old of both sexes
* Pre-existent severe chronic conditions (e.g. chronic liver or kidney disease, chronic obstructive pulmonary disease)
* Living outside of the surrounding catchment areas of the 6 healthcare centers.
* Women internationally displaced, without a permanent home or identified physical address.
* Women planning to move elsewhere in the following 2 years
* Women that do not provide a written Informed Consent.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the adherence to a healthy lifestyle score at 24 months | Baseline and 24 months
  The adherence to a healthy lifestyle will be measured by using a validated questionnaire for weight control in lifestyle-related diseases that compromise 14 questions, 12 regarding diet and 2 related to physical activity. Each question has 5 multiple choice answers (A, B, C, D, E). This questionnaire provides a final score ranging between 14-65 points. A lower score indicates poor adherence to a healthy lifestyle, while a high score indicates good adherence.
Change from baseline in the adherence to a healthy lifestyle score at 12 months | Baseline and 12 months
  The adherence to a healthy lifestyle will be measured by using a validated questionnaire for weight control in lifestyle-related diseases that compromise 14 questions, 12 regarding diet and 2 related to physical activity. Each question has 5 multiple choice answers (A, B, C, D, E). This questionnaire provides a final score ranging between 14-65 points. A lower score indicates poor adherence to a healthy lifestyle, while a high score indicates good adherence.

SECONDARY OUTCOMES:
Change from baseline in the minimum diet diversity of women (MDD-W) questionnaire at 24 months | Baseline and 24 months
  The MDD-W dichotomous questionnaire developed by the Food and Agriculture Organization of the United Nations (FAO) will be used to measure women's diet diversity.
Change from baseline in the minimum diet diversity of women (MDD-W) questionnaire at 12 months | Baseline and 12 months
  The MDD-W dichotomous questionnaire developed by the Food and Agriculture Organization of the United Nations (FAO) will be used to measure women's diet diversity.
Change from baseline in the International Physical Activity Questionnaire at 24 months | Baseline and 24 months
  The International Physical activity Questionnaire (IPAQ) short Form will be used to assess the level of physical activity of the participants.
Change from baseline in the International Physical Activity Questionnaire at 12 months | Baseline and 12 months
  The International Physical activity Questionnaire (IPAQ) short Form will be used to assess the level of physical activity of the participants.
Change from baseline in weight at 24 months | Baseline and 24 months
  Weight will be measured in kg and by using a digital weight scale. The WHO STEPwise guideline will be followed for this measurement.
Change from baseline in weight at 12 months | Baseline and 12 months
  Weight will be measured in kg and by using a digital weight scale. The WHO STEPwise guideline will be followed for this measurement.
Change from baseline in Body mass index (BMI) at 24 months | Baseline and 24 months
  BMI will be calculated by using the formula BMI= weight in kg/height in meters squared.
Change from baseline in Body mass index (BMI) at 12 months | Baseline and 12 months
  BMI will be calculated by using the formula BMI= weight in kg/height in meters squared.
Change from baseline in waist circumference at 24 months | Baseline and 24 months
  Waist circumference will be measured in cm and y using a constant tension tape. The WHO STEPwise guideline will be followed for this measurement.
Change from baseline in waist circumference at 12 months | Baseline and 12 months
  Waist circumference will be measured in cm and y using a constant tension tape. The WHO STEPwise guideline will be followed for this measurement.
Change from baseline in glycemia at 24 months | Baseline and 24 months
  Glycemia will be measured in mg/dL by using by pricking the fingertip with a lancet and glucometer. The WHO STEPwise guideline will be followed for this measurement.
Change from baseline in glycemia at 12 months | Baseline and 12 months
  Glycemia will be measured in mg/dL by using by pricking the fingertip with a lancet and glucometer. The WHO STEPwise guideline will be followed for this measurement.
Change from baseline in systolic and diastolic blood pressure at 24 months | Baseline and 24 months
  Systolic and diastolic blood pressure will me measured in mm Hg and by using an OMRON. The WHO STEPwise guideline will be followed for this measurement.
Change from baseline in systolic and diastolic blood pressure at 12 months | Baseline and 12 months
  Systolic and diastolic blood pressure will me measured in mm Hg and by using an OMRON. The WHO STEPwise guideline will be followed for this measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Jean C. Kalobu, MD; MPH, Principal Investigator — Memisa; José L. Peñalvo, PhD, Principal Investigator — Institute of Tropical Medicine; Diana M. Sagastume, MSc, Principal Investigator — Institute of Tropical Medicine
Locations (6):
- Democratic Republic of the Congo (6):
  - KAVWAYA, Kisantu, Bas-Congo Province
  - KINKOKA, Kisantu, Bas-Congo Province
  - MADIMBA, Kisantu, Bas-Congo Province
  - NGEBA, Kisantu, Bas-Congo Province
  - NKANDU 1, Kisantu, Bas-Congo Province
  - Kintanu Etat, Kisantu, Kongo Cnetral

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sagastume D, Sibongwere DK, Kidima O, Kembo DM, N'keto JM, Dimbelolo JC, Nkakirande DB, Kabundi JCK, Penalvo JL. Improving lifestyle behaviours among women in Kisantu, the Democratic Republic of the Congo: A protocol of a cluster randomised controlled trial. PLoS One. 2022 Sep 9;17(9):e0274517. doi: 10.1371/journal.pone.0274517. eCollection 2022. PMID 36084047
- See also: Improving lifestyle behaviours among women in Kisantu, the Democratic Republic of the Congo: A protocol of a cluster randomised controlled trial — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0274517